CLINICAL TRIAL: NCT06605651
Title: A Phase II Proof of Concept Multicenter, Randomized, Double-Blind Study to Assess the Safety and Efficacy of Phage Therapy in Patients with Hip or Knee Prosthetic Joint Infection Due to Staphylococcus Aureus Treated by DAIR
Brief Title: Proof of Concept Study to Assess Safety and Efficacy of Phage Therapy in Hip or Knee Prosthetic Joint Infections Due to Staphylococcus Aureus Treated by DAIR.
Acronym: GLORIA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Phaxiam Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PP-SA-003; 2024-516555-40-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-29; First posted 2024-09-20 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Hip Prosthesis Infection; Knee Prosthesis Infection
Keywords: Prosthetic Joint Infection; PJI; Bacteriophages; Phages; DAIR; Phage Therapy; Antimicrobials
MeSH Terms: interventions — Injections, Intra-Articular; Saline Solution

STUDY DESIGN:
Intervention Model Description: This is an international, multicentric, phase II (proof of concept), randomized, double-blind, parallel group, placebo-controlled study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study personnel (Investigator and their team, Sponsor's and CRO's Clinical Study Team will be blinded to subject treatment assignments except for the investigational pharmacist at each study site.
  The IWRS system will keep a coding list identifying the randomization number and the nature of the treatment allocated to each randomized patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Arm (Experimental): Anti-Staphylococcus aureus Bacteriophages (PP1493 and PP1815) intra-articular injection with 0.9% NaCl solution
  Interventions: Biological: Anti-Staphylococcus aureus Bacteriophages (PP1493 and PP1815) intra-articular injection with 0.9% NaCl solution
- Control Arm (Placebo Comparator): 0.9% NaCl solution
  Interventions: Drug: 0.9% NaCl solution

INTERVENTIONS:
Biological: Anti-Staphylococcus aureus Bacteriophages (PP1493 and PP1815) intra-articular injection with 0.9% NaCl solution — Three intra-articular injections during and/or following DAIR procedure
  Arms: Active Arm
Drug: 0.9% NaCl solution — Three intra-articular injections during and/or following DAIR procedure
  Arms: Control Arm

SUMMARY:
Total joint replacements are effective for chronic pain but can lead to Prosthetic Joint Infections (PJI), primarily caused by Staphylococcus aureus and resistant to antibiotics. Standard treatment involves DAIR surgery and antibiotics, but there's a need for better solutions due to rising infections and antibiotic resistance. Bacteriophage therapy, which targets specific bacteria, shows promise. Phaxiam Therapeutics is studying the safety and efficacy of phage therapy in treating Staphylococcus aureus infections in hip or knee PJI patients undergoing DAIR.

DETAILED DESCRIPTION:
Total joint replacement serves as valuable interventions in the management of chronic refractory pain when the other conservative treatments have not worked. They play a vital role in alleviating discomfort and improving the quality of life of subjects battling with joint diseases. However, the joint replacements present the challenge of Prosthetic Joint Infection (PJI). PJI have serious complications and can lead to significant mortality, morbidity, and healthcare expenditure.

The leading cause of PJI is gram-positive cocci, specifically Staphylococcus aureus. Bacterial biofilms, mainly formed with Staphylococcus, represent a significant challenge in the treatment of PJIs due to their resistance to antibiotic therapy. Standard of Care (SOC) for these complex infections is characterized primarily by an initial surgery (Debridment Antibiotics and Implant Retention (DAIR) and various regiments and combinations of antibiotics. While the patterns of utilization vary between institutions and geography, DAIR is considered low-invasive procedure, characterized by the possibility of not explanting the prosthetic implant and resecting the bone. The growing demand for joint arthroplasty and current PJI rates, combined with antibacterial resistance, clearly indicate an unmet medical need in treating biofilm-based PJIs.

Bacteriophage therapy could potentially improve the treatment paradigm for PJIs. Bacteriophages naturally occur with highly specific bacterial viruses that infiltrate bacterial cells, disrupting their metabolism, and causing bacterial lysis. Initial in vivo studies of phage therapy for bone-related infections have shown promise.

Phaxiam Therapeutics, a biotechnology company specializing in the research and development of anti-infective therapies using bacteriophages., has collections of phages against Escherichia coli, Pseudomonas aeruginosa, and Staphylococcus aureus. These phages have shown promise in preliminary tests and studies.

The objective of GLORIA study Is to assess the safety and efficacy of phage therapy versus placebo in treating Staphylococcus aureus infections in hip or knee PJI patients undergoing DAIR.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years
2. Knee or Hip PJI according to EBJIS (European Bone and Joint Infection) or ICM (International Consensus Meeting) guidelines
3. Monobacterial Infection due to S. aureus
4. Without preoperative diagnosis of superinfection due to another pathogen if treatment is administered at the end of the DAIR (presence of a contaminant is not considered clinically relevant)
5. Without diagnosis of superinfection due to another pathogen identified within 72h after bacteriological sample performed during the DAIR if treatment is administered up to 14 days after the DAIR
6. Indication for Open DAIR decided by the Multidisciplinary Team and/or Principal Investigator
7. S. aureus in joint fluid during the pre-inclusion period or in case of relapse of infection under antibiotics therapy in the last 6 months before inclusion
8. Patient with a life expectancy of 1 year or more as determined by the principal investigator.
9. Females of childbearing potential/Sexually active males with partner of childbearing potential: commitment to consistently and correctly use an acceptable effective method of birth control until 1 month after the last study drug administration.
10. Females of non-childbearing potential: either surgically sterilized or at least 1 year postmenopausal (amenorrhea duration at least 12 months)

Exclusion Criteria:

1. Relapse between DAIR and study drug administration planned up to 14 days after the DAIR.
2. Patients who have two planned DAIR in sequence (double DAIR)
3. Patients with ASA score ≥ 4
4. Severe sepsis or Septic shock or hemodynamic instability
5. Patients with an indication for fixed prosthesis exchange, or for joint fusion or for amputation
6. Indication for suppressive antibiotherapy
7. Immunosuppressed patients: Patients having a weakened immune system due to diseases conditions (i.e. genetic disorders, malnutrition) or treatment (i.e. anticancer drugs or organ transplant)
8. Positive Human Immunodeficiency Viruses (HIV) test or active hepatitis B and C
9. Previous treatment by bacteriophages
10. Any known phage allergy and/or to its excipients
11. Elevated ALT or AST above 4 times ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of phage therapy + DAIR compared with placebo + DAIR | From enrollment up to 3 months
  Incidence of serious adverse events
To assess the efficacy of phage therapy + DAIR compared with placebo + DAIR | From enrollment up to 3 months
  Percentage of patients with clinical cure

SECONDARY OUTCOMES:
To assess the safety of phage therapy + DAIR compared with placebo + DAIR | From enrollment up to 12 months
  Incidence of all adverse events and all safety parameters
To assess the efficacy of phage therapy + DAIR compared with placebo + DAIR | From enrollment up to 12 months
  Percentage of Patient with clinical cure from S.aureus's infection up to 6 months and up to 12 months. Percentage of patients with relapse exclusively due to another germ than Staphylococcus aureus up to 3 months, 6 months and 12 months
To describe the immunological response in serum and in joint fluid | From enrollment up to 3 months
  Titration of anti-Staphylococcus aureus phage antibodies
To describe the S. aureus bacterial load (bacteriology) in the joint fluid up to 1 month | From enrollment up to 1 month
  Quantitative or Semi-Quantitative analysis of bacterial load
To describe Cytology in the joint fluid | From enrollment up to 1 month
  Quantification and identification of polynuclear of joint fluid
To describe the hospitalization duration | From enrollment up to 3 months and up to 12 months
  Number of hospitalizations
To describe the hospitalization duration | From enrollment up to 3 months and up to 12 months
  Total duration of hospitalizations
To describe the quality of life for patients | From enrollment up to 3 months and up to 12 months
  Results of quality-of-life questionnaires (EQ-5D-5L: EuroQol-5 Dimensions-5 Levels) from 0 (worst health you can imagine) to 100 (best health you can imagine)
To describe joint function rehabilitation | From enrollment up to 3 months and up to 12 months
  Total score of either KOOS-12 (Knee Injury and Osteoarthritis Outcome Score 12 questions) OR HOOS-12 (Hip Injury and Osteoarthritis Outcome Score-12 questions) Questionnaires, depending on infected joint. The score is calculated in a scale from 0 (extreme symptoms) to 100 (absence of symptoms).
To describe the evolution of the prosthetic joint infection by X Ray image | From screening up to 3 months and up to 12 months
  X Ray image analysis to detect the potential appearance of abnormal loosening (border with shifting of the prosthesis)

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Chief Medical Officer, Study Director — Phaxiam Therapeutics; Audrey Study Team Leader, Study Director — Phaxiam Therapeutics

IPD SHARING:
Plan to Share IPD: No